CLINICAL TRIAL: NCT03213951
Title: Pilot Ex-Vivo Investigation of an Experimental Beta Probe for Assessment and Guidance of Prostate Cancer Resection
Brief Title: Ex-vivo Investigation of Beta Probe for Prostate Cancer Resection and Evaluation of PSMA-PET for Diagnosis of Intraprostatic Lesions
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: IntraMedical Imaging, LLC (Unknown)
Responsible Party: Principal Investigator, Clinton Bahler, Assistant Professor of Medicine, Indiana University
Other Study IDs: IUSCC-0615
Record Dates: First submitted 2017-07-08; First posted 2017-07-11 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: Surgical resection; Margins of resection; Beta radiopharmaceutical; Beta probe device; Ex-vivo
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate cancer: Gleason grade group 1-5 on prostate biopsy or prostate cancer recurrence.
  Interventions: Other: Experimental beta probe; Diagnostic Test: PSMA-PET

INTERVENTIONS:
Other: Experimental beta probe — 3mCi (or similar) dose of 68Ga-PSMA-11 will be given prior to resection of cancer. Experimental beta probe designed to detect 68Ga-PSMA-11 will be used on prostate tissue after it has been surgically removed.
Diagnostic Test: PSMA-PET — PSMA-PET imaging done prior to surgery and compared to whole mount imaging.

SUMMARY:
68Ga-PSMA is a radiopharmaceutical used with PET imaging for the detection of prostate cancer under a compassionate IND in patients who have presented with biochemical failure. In this study, the use of 68Ga-PSMA-11 will be extended to newly diagnosed patients with high risk prostate cancer. Patients enrolled to this study will undergo a 68Ga-PSMA-11 PET/CT or PET/MRI scan for research purposes (in addition to the routine CT or MRI that is routinely done for staging), and a second 68Ga-PSMA-11 administration just prior to surgery for experimental ex-vivo beta probe testing of resected tissue. Immediately following resection of the prostate, the intact tissue will be scanned using a PET camera designed for animal research in order to record the 68Ga-PSMA-11 distribution in the isolated tissue at higher resolution than can be attained using whole-body PET imaging. The experimental beta probe will then be use to measure 68Ga-PSMA-11 counts of the resected tissue.

DETAILED DESCRIPTION:
Primary Objective To assess beta ray detection of prostate cancer ex-vivo using experimental beta probe immediately after prostate cancer removal as determined by pathologist.

Secondary Objectives

* Compare preoperative standard of care staging via CT or MRI to 68Ga-PSMA-11 PET (CT or MRI) findings.
* Compare preoperative 68Ga-PSMA-11 PET (CT or MRI) lesion measurements with postoperative high-resolution PET of ex-vivo tissue.
* To compare the findings of each of the 68Ga-PSMA-11 detection methods to the surgical observations and the clinical tissue histopathology findings.

Exploratory Objective Correlation of beta probe measurements with preoperative 68Ga-PSMA-11 PET (CT or MRI) lesion measurements, postoperative PET/CT ex-vivo images, surgical observations, and pathology findings.

ELIGIBILITY:
Inclusion Criteria

To be considered eligible to participate in this study, a patient must meet all the inclusion criteria listed below:

1. ≥ 18 years of age
2. Must provide written informed consent
3. Presence of high grade prostate cancer (Gleason grade group 1-5) on prostate biopsy or prostate cancer recurrence.
4. Scheduled for prostate cancer removal
5. Willing and able to lie still for approximately 30 minutes in an enclosed space for the 68Ga-PSMA-11 PET CT or MRI

Exclusion Criteria

1. Participation in another investigational trial involving research exposure to ionizing radiation concurrently or within 30 days.
2. Significant acute or chronic medical, neurologic, or psychiatric illness in the subject that, in the judgment of the Principal Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This patient population will have Prostate cancer with planned surgical resection (GG2-5) of prostate cancer as part of routine clinical care or active surveillance/HIFU (GG1-3).
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Proportion of patients where prostate cancer was detected using the beta probe on excised prostate tissue | 1 day

SECONDARY OUTCOMES:
Proportion of patients who had cancer detected by both the standard of care imaging (CT or MRI) and the 68Ga-PSMA-11 PET (CT or MRI) imaging | 1 day
Proportion of patients who had cancer detected by the beta probe on excised prostate tissue compared with surgical observations | 1 day
Proportion of patients who had cancer detected by the beta probe on excised prostate tissue compared with clinical tissue histopathology observations | 1 day
Comparison of pre-operative 68Ga-PSMA-11 (CT or MRI) lesions measurements with post-operative ex-vivo PET of prostate tissue | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Clinton D. Bahler, MD, MS, Principal Investigator — Indiana Unversity
Locations (2):
- United States (2):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bahler CD, Green M, Hutchins GD, Cheng L, Magers MJ, Fletcher J, Koch MO. Prostate Specific Membrane Antigen Targeted Positron Emission Tomography of Primary Prostate Cancer: Assessing Accuracy with Whole Mount Pathology. J Urol. 2020 Jan;203(1):92-99. doi: 10.1097/JU.0000000000000501. Epub 2019 Aug 20. PMID 31430234